CLINICAL TRIAL: NCT03914651
Title: Comparison of Cumulative Live Birth Rate Per Initial Cycle Between 300 IU and 150IU Starting Dose of rFSH Among Aged Patients With Poor Ovarian Reservation: a Randomized Controlled Trail
Brief Title: CLBR Per Initial Cycle With Different Starting Dose in Aged Patients With Poor Ovarian Reservation: 300IU Versus 150IU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019002
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 300IU rFSH stimulation group (Active Comparator): 300IU rFSH stimulation group is defined as patients using gonadotropin-releasing hormone（GnRH）antagonist protocol with a 300IU rFSH Gonal-F® starting dose during controlled ovarian stimulation.
  Interventions: Drug: 300IU rFSH Gonal-F® starting dose during controlled ovarian stimulation
- 150IU rFSH stimulation group (Experimental): 150IU rFSH Gonal-F® stimulation group is defined as patients using GnRH antagonist protocol with a 150IU rFSH starting dose during controlled ovarian stimulation.
  Interventions: Drug: 150IU rFSH Gonal-F® starting dose during controlled ovarian stimulation

INTERVENTIONS:
Drug: 300IU rFSH Gonal-F® starting dose during controlled ovarian stimulation — On menstrual cycle day 2 or day 3, 300IU rFSH Gonal-F® will be administrated daily till the day of trigger. The dosage of rFSH can be adjusted only if there is a risk of ovarian hyperstimulation syndrome（OHSS）.
  Arms: 300IU rFSH stimulation group
Drug: 150IU rFSH Gonal-F® starting dose during controlled ovarian stimulation — On menstrual cycle day 2 or day 3, 150IU rFSH Gonal-F® will be administrated daily till the day of trigger. The dosage of rFSH can be adjusted only if there is a risk of OHSS or insufficient follicular growth.
  Arms: 150IU rFSH stimulation group

SUMMARY:
Among aged patients with poor ovarian reservation(defined as age 35 to 42 years; antral follicle count（AFC）≤ 5 or anti-mullerian hormone（AMH）≤ 1.2 ng/ml), cumulative live birth rate(CLBR) and time to live birth(TTLB) of the first stimulation cycle were compared between a starting dose of 300IU or 150IU rFSH in controlled ovarian stimulation with gonadotropin-releasing hormone（GnRH）antagonist protocol. This study is a prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age Limits≥35 and≤42；
2. AFC≤5 or AMH≤1.2ng/ml；
3. BMI≤30kg/m2；
4. The first IVF/intracytoplasmic sperm injection （ICSI） cycle；

Exclusion Criteria:

1. Any other underlying disease or condition considered IVF is contraindicated.
2. Ovarian hyperstimulation syndrome（PCOS）, moderate or severe intrauterine adhesion，untreated hydrosalpinx, adenomyosis， any myoma in cases that endometrium was affected, intramural larger than 4cm.
3. Autoimmune antibody positive, untreated.
4. History of recurrent miscarriages.
5. Patients seeking for Preimplantation Genetic Testing(PGT) treatment.
6. Simultaneous participation in another clinical study.
7. According to the judgment of the investigator, any reason or condition that precludes subject for participating in the study.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 22 months
  Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation after our interventions。And cumulative live birth rate is calculated by dividing the number of women achieving live birth after transfers of all study-specific embryos (within 1 year after randomization) by the total number of women randomized to the specific group.

SECONDARY OUTCOMES:
Time to live birth | 22 months
  Time to live birth is defined as the interval between the date of randomization and achieving live birth.
Cycle cancellation rate | 1 month
  Cycle cancellation is defined as cycle cancelled before obtaining at least one viable embryo for any reason. And cycle cancellation rate is calculated by dividing the number of women cancelled their cycle before obtaining at least one viable embryo for any reason by the total number of women randomized to the specific group.
Number of MII eggs | 1 month
  MII eggs is defined as eggs retrieved that reach the MII phase.
Cumulative Clinic pregnancy rate | 14 months
  Clinic pregnancy will be diagnosed with the detection of an intrauterine gestation sac. And cumulative clinic pregnancy rate is calculated by the number of women who achieves clinical pregnancy after transfers of all study-specific embryos (within 1 year after randomization) by the total number of women randomized to the specific group.
cumulative pregnancy loss rate | 19 months
  Pregnancy loss is defined as a complete spontaneous abortion or a nonviable pregnancy before 28 weeks of gestation. And cumulative pregnancy loss rate is calculated as the number of pregnancy losses / number of clinical pregnancy after transfers of all study-specific embryos (within 1 year after randomization).
Implantation rate | 14 months
  Number of gestation sac detected / number of embryo transferred.
Multiple pregnancy rate | 22 months
  Number of multiple pregnancies / number of clinical pregnancies over (up to) 3 transfers within 1 year.
Neonatal malformation rate | 22 months
  Number of infant diagnosed as neonatal malformation / the total number of infant delivered after 28 weeks of gestation.
Good quality embryo rate | 1 month
  Good quality embryo is defined as embryo that is graded as 6CII or better or blastocyst. And good quality embryo rate is calculated by dividing the number of good quality embryo by the total number of embryo obtained after fertilization in the specific group.
Birth weight | 22 months
  Weight of newborns at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China